CLINICAL TRIAL: NCT05548179
Title: An In Depth Study Investigating The Experiences of Patients In Leiomyosarcoma Clinical Trials
Brief Title: Exploring Clinical Trial Experiences of People With Leiomyosarcoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 87688730
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2022-09

CONDITIONS: Leiomyosarcoma
Keywords: leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical study participation has historically been heavily biased toward specific demographics.

Several people will be invited to enroll in this study so that it may collect a variety of data about leiomyosarcoma clinical trial experiences and identify barriers to participation as well as the causes of participants' failure or withdrawal.

People with leiomyosarcoma who are invited to take part in medical research will benefit from the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Patient has self-identified as planning to enroll in an interventional clinical trial
* Patient has been diagnosed with leiomyosarcoma
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Patient does not understand, sign, and return consent form
* Inability to perform regular electronic reporting
* Patient is pregnant
* ECOG score of 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Leiomyosarcoma patients who are actively considering participating in an interventional clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in an leiomyosarcoma clinical trial | 3 months
Rate of patients who remain in leiomyosarcoma clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kantidakis G, Litiere S, Neven A, Vinches M, Judson I, Schoffski P, Wardelmann E, Stacchiotti S, D'Ambrosio L, Marreaud S, van der Graaf WTA, Kasper B, Fiocco M, Gelderblom H. Efficacy thresholds for clinical trials with advanced or metastatic leiomyosarcoma patients: A European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group meta-analysis based on a literature review for soft-tissue sarcomas. Eur J Cancer. 2021 Sep;154:253-268. doi: 10.1016/j.ejca.2021.06.025. Epub 2021 Jul 20. PMID 34298376
- [Background] Serrano C, George S. Leiomyosarcoma. Hematol Oncol Clin North Am. 2013 Oct;27(5):957-74. doi: 10.1016/j.hoc.2013.07.002. Epub 2013 Aug 26. PMID 24093170
- [Background] Kasper B, D'Ambrosio L, Davis EJ, Ingham M, Broto JM, Trent JC, van Houdt WJ, Van Tine BA. What Clinical Trials Are Needed for Treatment of Leiomyosarcoma? Curr Treat Options Oncol. 2022 Mar;23(3):439-449. doi: 10.1007/s11864-021-00928-y. Epub 2022 Mar 11. PMID 35275323

DOCUMENTS (1):
  • Informed Consent Form (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT05548179/ICF_000.pdf